CLINICAL TRIAL: NCT07301905
Title: Culturally Targeted Messaging and Parental Receptivity to the Human Papillomavirus Vaccine
Brief Title: Culturally Targeted Health Communication and Receptivity to the Human Papillomavirus Vaccine Among Parents in Flint, MI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Todd Lucas, Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 00630245
Record Dates: First submitted 2025-09-08; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: HPV Vaccination

STUDY DESIGN:
Intervention Model Description: This research will use a 2 (White, African American) x 3 (No message, Education-only message, Culturally targeted message) quasi-experimental design. All participants will be randomly assigned to a no-message control group or to receive educational materials about HPV vaccination. Half of African American parents who receive educational materials will also view culturally targeted messaging about the HPV vaccine.
Who Masked: Participant
Masking Description: Participants will be unaware of their assignment to a general, education-only versus culturally targeted messaging condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- African American Culturally Targeted Messaging (Experimental): Culturally targeted messaging about the HPV vaccine for African American parents
  Interventions: Behavioral: Culturally Targeted HPV Vaccine Health Messaging
- African American General, Education-Only Messaging (Active Comparator): African American participants receive general, education-only messaging about the HPV vaccine.
  Interventions: Behavioral: General HPV Vaccine Health Messaging
- African American No Message (No Intervention): African American participants receive no messaging about the HPV vaccine
- White General, Education-Only Messaging (Active Comparator): White participants receive general, education-only messaging about the HPV vaccine.
  Interventions: Behavioral: General HPV Vaccine Health Messaging
- White No Message (No Intervention): White participants receive no messaging about the HPV vaccine

INTERVENTIONS:
Behavioral: General HPV Vaccine Health Messaging — General, education-only messaging about the HPV vaccine does not include culturally targeted messaging.
  Arms: African American General, Education-Only Messaging; White General, Education-Only Messaging
Behavioral: Culturally Targeted HPV Vaccine Health Messaging — Educational messaging about the HPV vaccine includes culturally targeted messaging about the HPV vaccine.
  Arms: African American Culturally Targeted Messaging

SUMMARY:
The goal of this clinical trial is to learn if culturally targeted messaging about the human papillomavirus (HPV) increases receptivity to the HPV vaccine among African American parents of vaccine-eligible daughters. The main question it aims to answer is:

• Does culturally targeted messaging increase African American parents' intentions to vaccinate their daughter against HPV?

Research will compare culturally targeted messaging to general, educational messaging and no messaging.

Participants will:

* View culturally targeted messages, education-only messages, or no messages about the HPV vaccine
* Report their intentions to vaccinate their daughter against HPV
* Report whether they have initiated HPV vaccination for their daughter six months later

DETAILED DESCRIPTION:
Cervical cancer incidence and mortality are higher for African American women than for White women. The human papillomavirus (HPV) vaccine is the most effective strategy for reducing risk for cervical cancer. However, African American girls are less likely to have completed the HPV vaccine series than White girls. The present research will evaluate a culturally targeted approach to health messaging about the HPV vaccine for parents with vaccine-eligible daughters. The central hypothesis is that African American parents will have greater receptivity to the HPV vaccine after receiving culturally targeted messaging compared to parents who receive no messaging or education-only messaging about HPV vaccination. The primary aims are: 1) evaluate effects of HPV vaccine education on White and African American parents' receptivity to the HPV vaccine, and whether culturally targeted messaging enhances HPV vaccine receptivity among African American parents, 2) compare effects of education-only versus culturally targeted messaging on activation of racism-related thinking when considering child HPV vaccination, and 3) examine the effects of racism-related medical mistrust on the effectiveness of culturally targeted messaging. General and culturally targeted messaging about the HPV vaccine were developed in collaboration with community members and a local health educator. Participants will report their intentions to vaccinate their daughter against HPV immediately after viewing health messaging, as well as initiation of the HPV vaccine series for their daughter 6-months post-messaging.

ELIGIBILITY:
Inclusion Criteria:

* Identify as Black/African American or White/Caucasian
* Have at least one daughter who is between 8-17 years of age, who is not currently pregnant, and who has not received any doses of the HPV vaccine

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 265 (Estimated)
Dates: Start 2024-11-17 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
HPV Vaccine Attitudes | Immediately following and 6-months post-health messaging
  Subscale of Theory of Planned Behavior measuring attitudes toward the HPV vaccine on response scale ranging from 1 = Strongly disagree to 7 = Strongly agree, where higher average scores indicate more positive attitudes
HPV Vaccine Normative Beliefs | Immediately following and 6-months post-health messaging
  Subscale of Theory of Planned Behavior measuring the extent to which participants believe other people are favorable toward the HPV vaccine on response scale ranging from 1 = Strongly disagree to 7 = Strongly agree, where higher average scores indicate stronger normative beliefs
HPV Vaccine Perceived Behavioral Control | Immediately following and 6-months post-health messaging
  Subscale of Theory of Planned Behavior measuring beliefs about ability to vaccinate their child on response scale ranging from 1 = Strongly disagree to 7 = Strongly agree, where higher average scores indicate greater perceived behavioral control
HPV Vaccine Intentions | Immediately following and 6-months post-health messaging
  Subscale of Theory of Planned Behavior measuring intentions to vaccinate their child on response scale ranging from 1 = Strongly disagree to 7 = Strongly agree, where higher average scores indicate greater intentions
Vaccination Initiation | 6-months post-health messaging
  1 self-report item measuring whether parents' daughters have received at least one dose of the HPV vaccine since completion of the initial survey, with Yes/No response options
Vaccination Discussion | 6-months post-health messaging
  1 self-report item measuring whether parents have discussed the HPV vaccine with their daughters' healthcare provider since completion of the initial survey, with Yes/No response options

SECONDARY OUTCOMES:
Anticipatory Racism | Immediately following health messaging
  3 items measuring the extent to which parents expect racism-related factors to interfere with getting the HPV vaccine for their daughter on a 7-point response scale on response scale ranging from 1 = Strongly disagree to 7 = Strongly agree, where higher average scores indicate greater expectations of racism

CONTACTS AND LOCATIONS:
Locations (1):
- Flint Journal Building, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided